CLINICAL TRIAL: NCT04096092
Title: A Population PK Study Into Teicoplanin in Intensive Care and Haematology Patients - a Strategy Towards Model Informed Precision Dosing
Brief Title: Pharmacokinetics of Teicoplanin in Intensive Care and Haematology Patients
Acronym: PLATO
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF 19.05
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Bacterial Infections
Keywords: Teicoplanin; Pharmacokinetics; Critically ill
MeSH Terms: conditions — Bacterial Infections; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Characterize teicoplanin PK in critically ill patients with a specific focus on alterations of exposure due to variability in renal function.

In a prospective, observational, open-label study the investigators aim to define PK of free drug concentrations of teicoplanine in ICU and heamatology patients and define a PK model for Bayesian dose individualization.

DETAILED DESCRIPTION:
Bacterial infection with coagulase-negative staphylococci (CNS) or methicillin resistant and sensitive staphylococcus aureus(MRSA/MSSA) indicates poor prognosis and increased mortality in critically ill patients.

With the current emergence of glycopeptide-intermediate sensitive Staphylococcus aureus strains, personalized dosing of teicoplanin is of utmost importance to preserve the current therapeutic armamentarium.

Teicoplanin is considered equipotent to vancomycin, albeit safer with minimal nephrotoxicity. It is estimated that 50% of all critically ill patients treated with teicoplanin does not reach target exposure. This is the major driver for treatment failure and development of resistance and dose individualization will overcome this problem.

Our project is aimed at developing and implementing a personalized dosing strategy for teicoplanin, to prevent development of glycopeptide resistance and allow safe treatment of glycopeptide intermediate sensitive bacteria.

In a prospective clinical study, critically ill patients (defined as ICU and hematology patients) who receive teicoplanin as standard care for antimicrobial treatment will be eligible for inclusion. Minimally invasive blood sampling for pharmacokinetic analysis will be retrieved through an indwelling central venous catheter or an arterial line (9 samples per patient). Teicoplanin total and free drug concentrations will be measured using a validated analytical assay. A total of 30 patients will be included.

We will develop a population PK model using nonlinear mixed effects modelling for total and unbound teicoplanin to characterize the magnitude of inter-individual variability in PK parameters (clearance, distribution volume), and to identify patient-derived characteristics that can predict such variability in a critically ill patient population.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is admitted to the ICU of the haematology department
2. The patient is at least 18 years of age on the day of inclusion
3. Is managed with a central venous catheter or arterial line
4. Is treated with teicoplanin as a part of standard care

Exclusion Criteria:

1. Has previously participated in this study
2. Patient is admitted to the haematology department and receives any form of RRT other than continuous venovenous hemofiltration (CVVH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill patients (defined as ICU and hematology patients) with a suspected or proven bacterial infection who are already treated with teicoplanin as a part of routine clinical care are eligible for inclusion. A total of 30 patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Total drug clearance | 4 days
  Pharmacokinetic curves will be taken

SECONDARY OUTCOMES:
Volume of distribution | 4 days
  Pharmacokinetic curves will be taken
Area under the curve | 4 days
  Pharmacokinetic curves will be taken

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided